CLINICAL TRIAL: NCT04709029
Title: Effect of Intravenous Versus Intrathecal Dexamethazone in Bupivacaine Spinal Anesthesia on Postdural Puncture Headache
Brief Title: Effect of Intravenous Versus Intrathecal Dexamethazone on Postdural Puncture Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Elsayed Elagamy, Assisstant professor Anesthesia,Intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 32/2020
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Postdural Puncture Headache
Keywords: intravenous dexamethazone; intrathecal dexamethazzone
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participant and outcome assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous dexamethazone group (Active Comparator): Patients receive intrathecal 3 ml heavy bupivacaine 0. 5% +1 ml normal saline + intravenous 8 mg dexamethazone in 10 ml saline,to prevent postdural puncture headache. Spinal anesthesia will be done in a sitting position under complete aseptic techniques, 25 G Quincke needle was inserted intrathecally at L3-L4 or L4-L5 interspace through midline approach. The study drugs were given by an anesthesiologist not aware of the type of medications injected.
  Interventions: Drug: Dexamethasone intravenous
- intrathecal dexamethazone group (Active Comparator): Patients receive intrathecal 3 ml heavy bupivacaine 0.5% + 4 mg (1 ml) dexamethazone + intravenous 10 ml normal saline to prevent postdural puncture headache. Spinal anesthesia will be done in a sitting position under complete aseptic techniques, 25 G Quincke needle was inserted intrathecally at L3-L4 or L4-L5 interspace through midline approach. The study drugs were given by an anesthesiologist not aware of the type of medications injected.
  Interventions: Drug: Dexamethasone intrathecal

INTERVENTIONS:
Drug: Dexamethasone intravenous — Evaluation of intravenous dexamethazone in prevention of postdural puncture headache
  Arms: intravenous dexamethazone group
Drug: Dexamethasone intrathecal — Evaluation of intrathecal dexamethazone in prevention of postdural puncture headache
  Arms: intrathecal dexamethazone group

SUMMARY:
This study will be conducted at Ain Shams University Hospital in Operating Theatre after ethical committe approval number (MS 32/ 2020). It is a prospective randomized controlled study will be done on patients undergoing lower abdominal and lower limb surgeries under spinal anethesia,Eligible patients will be randomized by computer system to one of two groups, either intravenous dexamethazzoe 8 mg with intrathecal heavy bupivacaine 0.5% or intrathecal 4mg dexamethazone with intrathecal heavy bupivacaine 0.5%. .

DETAILED DESCRIPTION:
Patients will be randomly divided into two equal groups: Group 1: patients receive intrathecal 3 ml bupivacaine 0. 5% +1 ml normal saline + intravenous 8 mg dexamethazone in 10 ml saline. Group 2: patients receive intrathecal 3 ml bupivacaine 0. 5% + 4 mg (1 ml) dexamethazone + intravenous 10 ml normal saline. Upon patients' arrival into the operating room, peripheral oxygen saturation (SPO2), ECG, pulse rate (PR), and systolic and diastolic blood pressures will be monitored one of the researchers and recorded every 5 minutes till the end of surgery. In a sitting position and with antiseptic techniques, 25 G Quincke needle was inserted intrathecally at L3-L4 or L4-L5 interspace through midline approach. The study drugs were given by an anesthesiologist not not aware of the type of medications injected. Subsequently, the patients were put in the supine position, and given oxygen 3 L/minutes by nasal prongs.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I or II undergoing lower limb surgeries under spinal anesthesia
* Patients ASAI or II undergoing lower abdominal surgeries under spinal anesthesia.

Exclusion Criteria:

* Emergency surgeries.
* Patients with uncompensated heart diseases.
* Patients with coagulopathy.
* Presence of infection at site of injection of spinal anesthesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
Prevention of postdural puncture headache | 48 hours after spinal anesthesia
  prevention of postdural puncture headache after spinal anesthesia in the first 48 hours postoperatively

SECONDARY OUTCOMES:
Duration of sensory block | 4 hours from injection of drug in subarachnoid space.
  Duration of sensory block after spinal anesthesia from injection of drug till regain of sensation at level of T10

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt